CLINICAL TRIAL: NCT06803836
Title: Inducible Nitric Oxide Synthase and Proinflammatory Cytokines in Periodontal Disease: Impact of Glycemic Control in T2DM
Brief Title: Inflammatory Response and Gingival iNOS Levels in Diabetic vs. Non-Diabetic Periodontitis Patients
Status: Completed | Type: Observational
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Sude Yildirim, Principal Investigator, Research Assistant, Ondokuz Mayıs University
Other Study IDs: DHF.061
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Periodontitis; Type 2 Diabetes; Glycemic Control
Keywords: periodontitis; diabetes; iNOS; glycemic control
MeSH Terms: conditions — Periodontitis; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Systemically Healthy Participants with Periodontitis: This group includes participants with periodontitis but without any systemic conditions such as diabetes. Periodontitis diagnosis is based on clinical attachment loss (CAL) and probing depth (PD) criteria.
- Systemically and Periodontally Healthy Participants: This group includes systemically and periodontally healthy participants. They serve as a control group to compare inflammatory biomarker levels under healthy conditions.
- Uncontrolled T2DM Participants with Periodontitis: Participants in this group have Type 2 diabetes mellitus (T2DM) with HbA1c levels >7 (uncontrolled diabetes) and periodontitis. Periodontal and systemic conditions were assessed.
- Controlled T2DM Participants with Periodontitis: This group includes participants with T2DM whose diabetes is well-controlled (HbA1c ≤7) and who have periodontitis. Clinical evaluations were performed.
- Controlled T2DM Periodontally Healthy Participants: Participants in this group have controlled T2DM (HbA1c ≤7) but no periodontal disease. They serve as a control group for comparing biomarker levels under controlled glycemic conditions.
- Uncontrolled T2DM Periodontally Healthy Participants: This group includes participants with uncontrolled T2DM (HbA1c >7) but no periodontal disease. Biomarker levels were measured to evaluate the effects of poor glycemic control on otherwise healthy periodontal tissues.

SUMMARY:
This study investigates the relationship between Type 2 diabetes mellitus (T2DM), glycemic control, and periodontal disease. Researchers analyzed the levels of inducible nitric oxide synthase (iNOS) and proinflammatory cytokines, such as tumor necrosis factor-alpha (TNF-α), interleukin-1 beta (IL-1β), and interferon-gamma (IFN-γ), in 118 participants. The participants were categorized based on their periodontal and diabetes control status.

DETAILED DESCRIPTION:
This study is an observational analysis using a cross-sectional time perspective and explores the interplay between Type 2 diabetes mellitus (T2DM), glycemic control, and periodontal disease by evaluating the expression of inducible nitric oxide synthase (iNOS) and proinflammatory mediators (TNF-α, IL-1β, IFN-γ, and PGE2) in gingival tissues. A total of 118 participants were classified into six groups based on their periodontal health and glycemic control status, determined by HbA1c levels.

Gingival biopsies were collected and analyzed using ELISA to measure biomarker levels. The study found significant differences in inflammatory marker concentrations between groups, with poorly controlled T2DM participants showing markedly higher levels of iNOS and cytokines. This aligns with the hypothesis that poor glycemic control amplifies periodontal inflammation and oxidative stress, contributing to tissue destruction.

The findings underline the critical role of glycemic regulation in managing periodontal disease and suggest potential targets, such as iNOS, for therapeutic interventions. This study adheres to ethical standards, including informed consent and approval by the Ondokuz Mayis University Clinical Research Ethics Committee. The results emphasize the bidirectional relationship between diabetes and periodontal health, contributing to a better understanding of the systemic implications of periodontal inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between 18 and 65 years of age (according to the World Health Organization definition of young and adult individuals).
* Diagnosed with periodontitis (Stage 2, 3, or 4) based on the 2017 Classification of Periodontal Diseases and Conditions.
* Diabetes control status determined by HbA1c levels: controlled diabetes: HbA1c ≤ 7, uncontrolled diabetes: HbA1c > 7
* Must volunteer and sign an informed consent form for clinical evaluations and collection of tissue samples.

Exclusion Criteria:

* History of smoking.
* Presence of systemic or local diseases affecting the immune system (e.g., autoimmune disorders, HIV, hepatitis).
* Pregnant or breastfeeding individuals.
* History of antibiotic use or periodontal treatment within the last 3-6 months.
* History of immunosuppressive therapy or chemotherapy.
* Requirement for antibiotic prophylaxis.
* Severe systemic illnesses unrelated to diabetes (e.g., cancer, cardiovascular diseases).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants will be selected from individuals seeking dental care at the Department of Periodontology, Faculty of Dentistry, Ondokuz Mayis University, Samsun, Turkey. The population includes adults with varying systemic and periodontal health statuses, such as individuals with Type 2 diabetes mellitus (T2DM) and/or periodontitis. Participants represent a diverse clinical population from the surrounding region and are recruited based on their suitability for the study's objectives.
Sampling Method: Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
Inducible Nitric Oxide Synthase (iNOS) concentration in gingival tissues | At baseline (single time point)
  iNOS levels will be measured in gingival tissue biopsies collected from all participants using ELISA. The aim is to assess the differences in iNOS expression across groups with varying periodontal and glycemic control statuses.

SECONDARY OUTCOMES:
Concentration of proinflammatory cytokines (e.g., TNF-α, IL-1β, IFN-γ, and PGE2) | At baseline (single time point)
  The levels of cytokines will be analyzed in gingival tissue samples to investigate their relationship with iNOS expression and differences between study groups.
Correlation between glycemic control (HbA1c levels) and iNOS/cytokine levels | At baseline (single time point)
  The study will examine the relationship between glycemic control (as determined by HbA1c levels) and biomarkers to evaluate the impact of diabetes control on periodontal inflammation.
Periodontal clinical parameters (e.g., probing depth, clinical attachment level) | At baseline (single time point)
  Clinical periodontal measurements, such as probing depth (PD) and clinical attachment level (CAL), will be recorded to assess the severity of periodontal disease in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Sude YILDIRIM BOLAT, DDS, Principal Investigator — Ondokuz Mayıs University, Department of Periodontology
Locations (1):
- Department of Periodontology, Faculty of Dentistry, Ondokuz Mayis University,, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The decision to not share individual participant data (IPD) is based on ethical considerations, institutional policies, and the need to protect participant privacy and confidentiality. The collected data will only be used for the purposes of this study and will not be made available for external use.